CLINICAL TRIAL: NCT04708093
Title: Effect of Whole Body Vibration Training on Selected Breast Cancer Risk Factors in Obese Postmenopausal Women: A Randomized Controlled Trial
Brief Title: Whole Body Vibration Training and Breast Cancer Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa A. Mohamed, Professor in Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Woman health
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hot Flashes; Prolactin; Whole Body Vibration
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Intervention Model Description: prospective study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration training (WBVT) (Experimental): whole body vibration group
  Interventions: Device: whole body vibration training
- Controlled (No Intervention): advised about healthy dieting

INTERVENTIONS:
Device: whole body vibration training — Oscillating platform
  Other Names: (WBVT)
  Arms: whole body vibration training (WBVT)

SUMMARY:
study aim is to determine the effect of whole body vibration training (WBVT) on body mass index, serum prolactin concentration as a risk factors for breast cancer and severity of hot flashes in obese postmenopausal women.

DETAILED DESCRIPTION:
Menopause is a physiological process characterized by spontaneous cessation of menstrual cycle lasting at least 12 months, it is normally occurring in women aged 45 - 55 years . Postmenopausal women have higher prevalence of menopausal symptoms that significantly affect their quality of life more than pre- and perimenopausal women .

Increased adiposity, as measured by high body mass index, is associated with more severe menopausal symptoms also, obese female has a high risk lifestyle for the development of post-menopausal breast cancer .

The link between BMI and breast cancer risk is likely to be due to increased concentrations of bioavailable estradiol, which results in turn from an increase in the production of estrogens by aromatase in the adipose tissue, conversion of hormones in fatty tissue and a decrease in the serum concentration. This is likely to explain the higher risk of breast cancer in overweight post-menopausal women .

Menopause is also associated with atherogenic changes, including a worsening of CVD risk factors and decreased aerobic fitness compared with premenopausal women.

This initially may be due to a decrease in endogenous estrogen levels, and likely further exacerbated by increased adiposity and reductions in exercise habits or physical activity levels.

Post menopausal women recorded a high serum prolactin concentration however, they have a significant chance of normalizing their prolactin levels.

Serum prolactin levels rise transiently after several physiological states including pregnancy, breast-feeding, exercise, meals, sexual intercourse, minor surgical procedures, general anesthesia, other forms of acute stress and menopause.

Estrogen is another key regulator of prolactin and has been shown to increase the production and secretion of prolactin from the pituitary gland. In addition to dopamine and estrogen, a whole range of other hormones can both increase and decrease the amount of prolactin released in the body, with some examples being thyrotropin-releasing hormone, oxytocin and anti-diuretic hormone .

Whole-body vibration training is a promising adjunct intervention therapy for management of obesity, as there is few evidence that it can reduces body mass index and enhances muscles strength.

In initial stage of obesity management, WBVT is highly recommended because it allows a mild joints stress, deconditioning for obese patient with poor motivation because it achieve its target without provoking an excessive fatigue. In addition, Passive vibrations do not involve voluntary movement and need a lower contribution of central command, so WBVT is as effective as aerobic and resistance exercise in reducing fat mass and moderating the deficit of the relative muscle strength . Lastly, WBVT may be effective in vascular health promotion and prevention in young obese women.

Whole body vibration training(WBVT) has been recognized as an effective alternative exercise modality to resistance exercise for its ability in enhancing force and power, generating capacity in skeletal muscle, increasing bone mass, improving cardiovascular function, reducing fat mass and moderating the deficit of the relative muscle strength. Unfortunately, the effect of resistance exercise on prolactin has not been extensively studied .

So, this study was conducted to evaluate the effect of whole body vibration training on BMI, waist circumference, serum prolactin concentration and hot flashes in obese postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* obese BMI ranged between 30-39.9 kg/m2.
* postmenopausal women

Exclusion Criteria:

* women with musculoskeletal or cardiovascular or neurological disorders
* hypothyroidism,
* polycystic ovary syndrome.
* chronic renal failure.
* participate in any exercise program prior to the study by six months.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — post menopausal female
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | after study completion through 3months
  kg\m2
serum prolactin concentration | after study completion through 3months
  ng\ml

SECONDARY OUTCOMES:
hot flashes | after study completion through 3months
  severity

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No